CLINICAL TRIAL: NCT00644085
Title: Does Low-Dose Aspirin Improve Outcome in IVF/ICSI? A Prospective, Randomized, Double Blind Placebo Controlled Trial
Brief Title: Does Low-Dose Aspirin Improve Outcome in In Vitro Fertilisation/Intra Cytoplasmatic Sperm Injection (IVF/ICSI)?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Kaatje Dirckx, MD, University Hospital Ghent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99/191
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Infertility
Keywords: IVF and ICSI
MeSH Terms: conditions — Infertility | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): oral administration of aspirin 100 mg
  Interventions: Drug: aspirin
- 2 (Placebo Comparator): oral administration of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aspirin — oral administration of aspirin 100 mg
  Arms: 1
Drug: placebo — oral administration of placebo
  Arms: 2

SUMMARY:
To investigate the effect of daily administration of low-dose aspirin, compared to placebo, on IVF and ICSI outcome.

ELIGIBILITY:
Inclusion Criteria:

* Dutch-speaking women
* Starting a first or second IVF/ICSI cycle

Exclusion Criteria:

* Women suffering from

  * platelet dysfunction
  * thrombopenia
  * gastro-intestinal ulcers
  * recurrent gastritis
  * aspirin hypersensitivity
* Women on treatment with anticoagulants or aspirin

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2000-04; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved
Clinical pregnancy rate per embryo transfer

SECONDARY OUTCOMES:
Live birth rate per cycle

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dhont, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Dirckx K, Cabri P, Merien A, Galajdova L, Gerris J, Dhont M, De Sutter P. Does low-dose aspirin improve pregnancy rate in IVF/ICSI? A randomized double-blind placebo controlled trial. Hum Reprod. 2009 Apr;24(4):856-60. doi: 10.1093/humrep/den476. Epub 2009 Jan 8. PMID 19131401
- See also: Related Info — http://www.uzgent.be